CLINICAL TRIAL: NCT06721195
Title: A Cross-Sectional Study on Euphoria Induced by Remimazolam During Gastrointestinal Endoscopy and Its Related Factors
Brief Title: Study on the Feelings of Euphoria Caused by Remimazolam During Gastroscopy and Colonoscopy and Their Related Factors
Acronym: ERGE
Status: Recruiting | Type: Observational
Sponsor: Zhangjie Yu (Other)
Responsible Party: Sponsor-Investigator, Zhangjie Yu, Attending Physician, RenJi Hospital
Organization: RenJi Hospital (Other)
Other Study IDs: LY2024-174-B
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Euphoria; Remimazolam Besylate; Gastrointestinal Endoscopy
MeSH Terms: interventions — remimazolam

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Remimazolam Sedation Group: his cohort includes patients undergoing painless gastrointestinal endoscopy (gastroscopy, colonoscopy, or both) who receive sedation with remimazolam. The study aims to evaluate the incidence of euphoria induced by remimazolam and explore related factors. All patients receive sedation according to standard clinical guidelines, including pre-procedural sufentanil and lidocaine gel for oral preparation, followed by remimazolam for induction and maintenance.
  Data collected include demographic characteristics, pre- and post-procedure euphoria scores assessed using the ARCI-MBG scale, perioperative safety indicators, and patient satisfaction.
  Interventions: Drug: Remimazolam for Gastrointestinal Endoscopy Sedation

INTERVENTIONS:
Drug: Remimazolam for Gastrointestinal Endoscopy Sedation — This intervention involves the use of remimazolam, a short-acting benzodiazepine, for sedation during gastrointestinal endoscopy procedures (gastroscopy, colonoscopy, or both). Remimazolam is administered intravenously at an initial dose of 0.2-0.3 mg/kg, followed by additional doses of 2.5 mg as needed to maintain adequate sedation (MOAA/S score ≤ 2).
  Unlike other benzodiazepines, remimazolam is rapidly metabolized by plasma esterases, resulting in a quick onset and recovery with minimal respiratory and cardiovascular depression. The study specifically evaluates the euphoria-inducing potential of remimazolam, using the ARCI-MBG scale pre- and post-procedure to assess its effect on patient comfort and satisfaction.

SUMMARY:
This study aims to investigate the incidence of euphoria induced by remimazolam during gastrointestinal endoscopy and explore its related factors. Gastrointestinal endoscopy, a minimally invasive procedure, often causes discomfort and anxiety for patients. Remimazolam, a short-acting benzodiazepine, is increasingly used for sedation during these procedures due to its rapid onset, short metabolism, and controlled cardiorespiratory effects. This cross-sectional study will evaluate the effect of remimazolam on patient comfort, cooperation, and satisfaction during endoscopy, aiming to optimize sedation protocols and improve clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years, regardless of gender.
* Patients scheduled for routine painless gastrointestinal endoscopy, including gastroscopy, colonoscopy, or both.
* ASA physical status classification: I or II.
* BMI between 18 kg/m² and 28 kg/m².
* Anticipated procedural duration of no more than 30 minutes.
* Patients who have provided written informed consent after understanding the study purpose, procedures, and potential risks.

Exclusion Criteria:

* History of psychiatric disorders such as schizophrenia, bipolar disorder, or personality disorders, or a history of alcohol, stimulant, or other substance abuse.
* Known allergies or intolerance to any medication used in the study, including remimazolam, sufentanil, or benzodiazepines.
* Patients requiring complex endoscopic procedures (e.g., ERCP, endoscopic submucosal dissection, endoscopic mucosal resection, or peroral endoscopic myotomy).
* History of severe hepatic or renal disease.
* Pregnant or lactating women.
* Participation in another clinical study within the past three months.
* Any condition or factor that, in the investigator's judgment, makes the patient unsuitable for participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients aged 18 to 65 years undergoing painless gastrointestinal endoscopy (gastroscopy, colonoscopy, or both) at a tertiary hospital. Participants must meet the inclusion criteria, such as ASA I-II classification and BMI between 18 and 28 kg/m². Patients are recruited from routine endoscopy appointments and provided written informed consent prior to participation. Exclusion criteria include severe comorbidities, psychiatric disorders, substance abuse, pregnancy, or recent participation in other clinical studies.
Sampling Method: Non-Probability Sample
Enrollment: 305 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Euphoria Induced by Remimazolam | From pre-procedure baseline to 2 hours post-procedure (Euphoria is assessed at two time points: immediately before sedation and two hours after the procedure, upon full recovery.)
  he occurrence of euphoria in patients undergoing sedation with remimazolam during gastrointestinal endoscopy procedures (gastroscopy, colonoscopy, or both). Euphoria is assessed using the ARCI-MBG scale. A positive result is defined as an increase in the ARCI-MBG score post-procedure compared to pre-procedure.

SECONDARY OUTCOMES:
factors Associated with Euphoria Induced by Remimazolam | From pre-procedure baseline to 2 hours post-procedure (Factors are collected before the procedure, during sedation, and 2 hours post-procedure, upon full recovery.)
  The identification of demographic, procedural, and clinical factors associated with the occurrence of euphoria induced by remimazolam during gastrointestinal endoscopy. Factors evaluated include age, gender, education level, BMI, ASA classification, comorbidities, dosage of remimazolam and sufentanil, procedural duration, perioperative adverse events, smoking and alcohol use, pre-procedural anxiety levels, and dream experiences.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared. Data will include demographic characteristics, procedural details, and outcome measures. Access will be granted to qualified researchers upon request via a secure data repository.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: De-identified individual participant data (IPD) will be available starting 6 months after the publication of the primary study results. Data will remain available for 5 years.
Access Criteria: Qualified researchers affiliated with academic, governmental, or non-profit institutions may request access to the IPD. Requests must include a detailed research proposal, institutional review board (IRB) approval (if applicable), and a signed data-sharing agreement. Access will be provided to de-identified data relevant to the study objectives, including demographic information, procedural details, and primary/secondary outcome measures. Data will be shared via a secure repository upon approval of the request.

REFERENCES:
- [Background] Basturk A, Artan R, Yilmaz A. Efficacy and safety of midazolam and ketamine in paediatric upper endoscopy. Arab J Gastroenterol. 2017 Jun;18(2):80-82. doi: 10.1016/j.ajg.2017.05.004. Epub 2017 Jun 1. PMID 28579345
- [Background] Brechmann T, Maier C, Kaisler M, Vollert J, Schmiegel W, Pak S, Scherbaum N, Rist F, Riphaus A. Propofol sedation during gastrointestinal endoscopy arouses euphoria in a large subset of patients. United European Gastroenterol J. 2018 May;6(4):536-546. doi: 10.1177/2050640617736231. Epub 2017 Oct 4. PMID 29881609
- [Background] Schippers F, Pesic M, Saunders R, Borkett K, Searle S, Webster L, Stoehr T. Randomized Crossover Trial to Compare Abuse Liability of Intravenous Remimazolam Versus Intravenous Midazolam and Placebo in Recreational Central Nervous System Depressant Users. J Clin Pharmacol. 2020 Sep;60(9):1189-1197. doi: 10.1002/jcph.1614. Epub 2020 Jun 3. PMID 32495449
- [Background] Ciraulo DA, Knapp CM, LoCastro J, Greenblatt DJ, Shader RI. A benzodiazepine mood effect scale: reliability and validity determined for alcohol-dependent subjects and adults with a parental history of alcoholism. Am J Drug Alcohol Abuse. 2001 May;27(2):339-47. doi: 10.1081/ada-100103713. PMID 11417943
- [Background] Tezcan AH, Ornek DH, Ozlu O, Baydar M, Yavuz N, Ozaslan NG, Dilek K, Keske A. Abuse potential assessment of propofol by its subjective effects after sedation. Pak J Med Sci. 2014 Nov-Dec;30(6):1247-52. doi: 10.12669/pjms.306.5811. PMID 25674117
- [Background] Zhao K, Yang N, Yue J, Han Y, Wang X, Kang N, Zhang T, Guo X, Xu M. Factors associated with euphoria in a large subset of cases using propofol sedation during gastrointestinal endoscopy. Front Psychiatry. 2023 Apr 27;14:1001626. doi: 10.3389/fpsyt.2023.1001626. eCollection 2023. PMID 37181900